CLINICAL TRIAL: NCT00977548
Title: Phase II Study Evaluating the Role of Erlotinib an Epidermal Growth Factor Receptor (EGFR) Inhibitor in the Treatment of Myelodysplastic Syndrome
Brief Title: Erlotinib Study for Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15961; OSI3666s (Other: Genentech)
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Results first posted 2013-09-16 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-05

CONDITIONS: Myelodysplastic Syndrome
Keywords: MDS; blood diseases; bone marrow; hematopoietic; leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Hematologic Diseases; Leukemia | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib Treatment (Experimental): Erlotinib was given as an oral 150 mg daily dose for 16 weeks. The dose was adjusted for diarrhea, rash and pulmonary toxicity.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Participants took erlotinib at least 1 hour before, or 2 hours after they ate a meal or snack. Participants were advised to take erlotinib at around the same time every day.
  Other Names: Tarceva; OSI-774

SUMMARY:
The purpose of this research study is to find out what effects, good and/or bad, erlotinib has on the patient and their myelodysplastic syndrome. Erlotinib has been approved by the Food and Drug Administration (FDA) to treat non-small cell lung cancer; however, erlotinib use in this study is considered investigational as the FDA has not approved it for the treatment of myelodysplastic syndrome.

DETAILED DESCRIPTION:
Screening Period: Informed consent, physical examination, medical history report, blood tests, pregnancy test (if applicable), list of current medications, description of symptoms, chest x-ray, ECG, bone marrow aspirate/biopsy within 4 weeks of study start.

Weeks 2,6,10 and 14: Blood tests.

Weeks 4 and 12: Blood tests, physical exam, patients will answer question about how they are feeling and if there are any changes to medication they have taken.

Weeks 8 and 16: Blood tests, physical exam, patients will answer question about how they are feeling and if there are any changes to medication they have taken, bone marrow aspirate/biopsy (if physician has determined the patient has had a clinical response or partial response to treatment.

After week 16 (if responding to treatment): Have a bone marrow aspirate/biopsy (will be repeated at time of relapse, i.e., more than 50% increase in the percentage of myeloblasts [leukemia cells] or drop in blood counts after they improved or requiring regular blood transfusions after not requiring them for at least 8 weeks, or after 1 year in study).

After the patient has stopped taking erlotinib: Periodic follow-up on patients' status.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have an established diagnosis of myelodysplastic syndrome (MDS) and have either: Low or intermediate 1 risk disease by International Prognostic Scoring System (IPSS) for MDS with symptomatic anemia (defined as hemoglobin less than 10.0 g/dl) or transfusion dependent anemia (defined as requiring ≥ 4 units of red blood cells (RBCs) administered with a pretreatment hemoglobin value of ≤ 9 g/dL in the 8 weeks prior to Day 1 of treatment in this study). Patients with anemia must have no response to at least to 6 weeks trial of erythroid stimulating agents (ESA) [erythropoietin/ darbepoetin]. Patients with serum erythropoietin levels more than 500 mU/ ml on diagnosis are eligible to the study without erythropoietin/darbepoetin prior treatment. Patients who do not meet anemia criteria are still eligible if they had thrombocytopenia with two or more platelet counts < 50 x 10^9/L or a significant clinical hemorrhage requiring platelet transfusions or if they had neutropenia with an absolute neutrophil count (ANC) < 1 x 10^9/L; Intermediate-2 or high risk MDS by IPSS.
* Patients ≥ 60 years with Acute Myeloid Leukemia (AML) by WHO classification and myeloblasts percentage 20-30% (RAEB-t by MDS French-American-British (FAB) classification) are eligible for the study if deemed not suitable for induction chemotherapy or declined that option.
* All prior treatment must have been discontinued 28 days prior to Day 1 of treatment in this study except (ESA) and colony stimulating factors where it should be stopped 14 days prior to start therapy on study, and hydroxyurea should be stopped 2 days before.
* Prior bone marrow or stem cell transplant is allowed.
* Secondary or therapy related MDS patients are eligible.
* Patients with chronic myelomonocytic leukemia (CMML) are eligible.
* Patients must have a performance status of 0 - 2 by Zubrod performance status criteria.
* Pretreatment pathology materials must be available for morphologic review. Collection of blood and marrow specimens for pathology review must be completed within 28 days prior to registration.
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for at least 2 years.
* In calculating days of tests and measurements, the day a test or measurement is done is considered Day 0. Therefore, if a test is done on a Monday, the Monday four weeks later would be considered Day 28. This allows for efficient patient scheduling without exceeding the guidelines. If Day 28 or 60 falls on a weekend or holiday, the limit may be extended to the next working day.
* All patients must be informed of the investigational nature of this study and must sign and give written consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Patients must not have received prior remission induction chemotherapy as treatment for MDS.
* Patients must not be pregnant or nursing because of the potential risks of the drugs used in this study. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Patients who are known HIV positive are not eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rami Komrokji, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2009 and January 2011, 39 patients signed consent at Moffitt Cancer Center.
Pre-assignment Details: 4 of the initial 39 patients were found to be ineligible after signing informed consent.
Period: Overall Study
Arm/Group | Erlotinib Treatment
Started | 39
Completed | 26
Not Completed | 13
Not completed — Ineligible | 4
Not completed — Adverse Event | 8
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 4 of the initial 39 patients were found to be ineligible after signing informed consent.
Arm/Group | Erlotinib Treatment
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 34
Age Continuous [Mean (Full Range); unit: years] | 73 [64 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Combined Overall Response Rate (ORR)
Description: Best Response Categories: Marrow complete response (CR), Bone marrow: ≤ 5% myeloblasts and decrease by ≥ 50% over pretreatment; Hematological improvement (HI), Hgb increase by ≥ 1.5 g/dL, Absolute increase of ≥ 30 x 10^9/L for patients starting with > 20 x 10^9/L, At least 100% increase and an absolute increase of > 0.5 x 10^9/L, as defined by the International Working Group (IWG) 2006 criteria.
Time Frame: Up to 21 Months
Population: All evaluable participants. Nine patients were not evaluable for response (withdrew consent or off study due to adverse event before first evaluation).
Measure: Number; unit: participants
Arm/Group | Erlotinib Treatment
Number analyzed (Participants) | 26
participants
  Marrow Complete Response (CR) | 3
  Hematological Improvement (HI) | 2
  Combined Overall Response | 5

2. Secondary Outcome: Median Overall Survival (OS)
Description: OS: The time from randomization until death from any cause. Kaplan-Meier estimates were used for secondary endpoint analysis.
Time Frame: Up to 21 Months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib Treatment
Number analyzed (Participants) | 26
months | 6.8 [4.9 to 13.2]

3. Secondary Outcome: Median Progression Free Survival (PFS)
Description: PFS: The time elapsed between treatment initiation and tumor progression or death from any cause. Kaplan-Meier estimates were used for secondary endpoint analysis. Disease Progression is defined using International Working Group (IWG) Response Criteria for MDS, as at least 50% decrement from maximum remission/response levels in granulocytes or platelets; reduction in hemoglobin (Hgb) concentration by ≥ 2 g/dL; transfusion dependence.
Time Frame: Up to 21 Months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib Treatment
Number analyzed (Participants) | 26
months | 3.6 [2 to 4.8]

4. Secondary Outcome: Leukemia Free Survival (LFS)
Description: LFS: Survival without evidence of relapse at any time post-transplant. Kaplan-Meier estimates were used for secondary endpoint analysis.
Time Frame: Up to 21 Months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib Treatment
Number analyzed (Participants) | 26
months | 5 [3.4 to 7.3]

ADVERSE EVENTS:
Time Frame: 1 year, 9 months
Arm/Group | Erlotinib Treatment
Serious Adverse Events (participants affected / at risk) | 24/35
Other Adverse Events (participants affected / at risk) | 32/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib Treatment (N=35)
Hemoglobin (Blood and lymphatic system disorders) | 10
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 5
Cardiac Arrhythmia - Other (Cardiac disorders) | 1
Cardiac ischemia/infarction (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 1
Coagulation - Other (Blood and lymphatic system disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 4
Fever (in the absence of neutropenia) (General disorders) | 2
Death not associated with CTCAE term - Death NOS (General disorders) | 3
Death not associated with CTCAE term - Disease progression NOS (General disorders) | 2
Death not associated with CTCAE term - Sudden death (General disorders) | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Anorexia (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 5
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1
Hemorrhage, CNS (Nervous system disorders) | 2
Hemorrhage, GI - Colon (Gastrointestinal disorders) | 2
Hemorrhage, GI - Lower GI NOS (Gastrointestinal disorders) | 1
Hemorrhage/Bleeding - Other (General disorders) | 1
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Abdomen NOS (Infections and infestations) | 1
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils -Blood (Infections and infestations) | 1
Infection (documented clinically or microbiologically) w/Grade 3 or 4 neutrophils - Lung (pneumonia) (Infections and infestations) | 2
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Mucosa (Infections and infestations) | 1
Infection - Other (Infections and infestations) | 8
Infection with normal ANC or Grade 1 or 2 neutrophils - Blood (Infections and infestations) | 3
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Sinus (Infections and infestations) | 1
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 1
Creatinine (Metabolism and nutrition disorders) | 1
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1
Mental status (Psychiatric disorders) | 1
Mood alteration - Depression (Psychiatric disorders) | 1
Neurology - Other (General disorders) | 2
Syncope (fainting) (General disorders) | 1
Pain - Abdomen NOS (General disorders) | 1
Pain - Back (General disorders) | 1
Pain - Chest wall (General disorders) | 1
Pain - Head/headache (General disorders) | 1
Pain - Other (General disorders) | 1
Pain - Throat/pharynx/larynx (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1
Renal failure (Renal and urinary disorders) | 3
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1
Vascular - Other (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib Treatment (N=35)
Diarrhea (Gastrointestinal disorders) | 23
Anorexia (Gastrointestinal disorders) | 14
Nausea (Gastrointestinal disorders) | 6
Gastrointestinal - Other (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 2
Pruritus/itching (Skin and subcutaneous tissue disorders) | 16
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 15
Dry skin (Skin and subcutaneous tissue disorders) | 9
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 8
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 2
Ulceration (Skin and subcutaneous tissue disorders) | 2
Fatigue (Asthenia, lethargy, malaise) (General disorders) | 17
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10^9/L) (General disorders) | 3
Sweating (diaphoresis) (General disorders) | 2
Weight loss (General disorders) | 2
Hemorrhage/Bleeding - Other (General disorders) | 6
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 4
Hemorrhage, GI - Colon (Gastrointestinal disorders) | 2
Hemorrhage, GI - Lower GI NOS (Gastrointestinal disorders) | 2
Infection - Other (Infections and infestations) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Blood (Infections and infestations) | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Eye NOS (Infections and infestations) | 2
Pain - Chest/thorax NOS (General disorders) | 2
Pain - Other (General disorders) | 2
Pain - Scalp (General disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7
Dizziness (General disorders) | 4
Platelets (Blood and lymphatic system disorders) | 4
Hemoglobin (Blood and lymphatic system disorders) | 2
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2
Edema: limb (Blood and lymphatic system disorders) | 2
Lymphatics - Other (Blood and lymphatic system disorders) | 2
Dry eye syndrome (Eye disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes